CLINICAL TRIAL: NCT01744288
Title: A Open Label, Randomized, Crossover and Potential Parallel, Single Dose Study of Ticagrelor 180 mg and Acetylsalicylic Acid (ASA) in Healthy Volunteers Followed by Autologous in Vivo Platelet Transfusion to Determine the Effects of Platelet Supplementation on the Reversibility of Platelet Inhibition
Brief Title: Study to See if Platelet Transfusion Stop or Lessen the Effect of the Drug on Platelets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D5130C00079
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Inhibition on Platelet Aggregation
Keywords: Phase 1 Safety ,; pharmacodynamic,; Ticagrelor,; Clopidogrel,; Platelets
MeSH Terms: interventions — Ticagrelor; Clopidogrel

ARMS (4):
- 1 (Experimental): Ticagrelor with Platelet transfusion
  Interventions: Drug: Ticagrelor; Drug: ASA
- 2 (Experimental): Ticagrelor without Platelet transfusion
  Interventions: Drug: Ticagrelor; Drug: ASA
- 3 (Active Comparator): Clopidogrel with Platelet transfusion
  Interventions: Drug: Clopidogrel; Drug: ASA
- 4 (Active Comparator): Clopidogrel without Platelet transfusion
  Interventions: Drug: Clopidogrel; Drug: ASA

INTERVENTIONS:
Drug: Ticagrelor — Oral single loading dose 180ng
  Arms: 1; 2
Drug: Clopidogrel — Oral single loading dose 600mg
  Arms: 3; 4
Drug: ASA — 81mg once daily from day -2 up to platelet transfusion

SUMMARY:
Study to see if platelet transfusion stop or lessen the effect of the drug on platelets

DETAILED DESCRIPTION:
A open label, randomized, crossover and potential parallel, single dose study of ticagrelor 180 mg and acetylsalicylic acid (ASA) in healthy volunteers followed by autologous in vivo platelet transfusion to determine the effects of platelet supplementation on the reversibility of platelet inhibition

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Healthy male and/or female volunteers aged 18 to 50 years, inclusive, with suitable veins for cannulation or repeated venipuncture. (Healthy as determined by medical history and physical examination, laboratory parameters, electrocardiogram (ECG) perform
* Have a body mass index (BMI) between 18 and 35 kg/m2 (inclusive) and weigh at least 50 kg and no more than 120 kg

Exclusion Criteria:

* ADP induced platelet aggregation <60% prior to platelet apheresis
* History of peptic ulcer disease Healthy volunteers with a propensity to bleed (eg, due to recent trauma, recent surgery, active or recent gastrointestinal bleeding or moderate hepatic impairment)
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of the investigational product
* Current smokers, those who have smoked or used nicotine products within the previous 3 months and those who tested positive for cotinine at screening or at admission to the study center

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 258 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics in terms of percent of inhibition of adenosine phosphatase (ADP)-induced platelet aggregation assessed by light transmission aggregometry (LTA) after loading dose of Ticagrelor | Predose, 0h, 2h,6h,12h,24h,36h,48h,60h,72h,84h and 96h

SECONDARY OUTCOMES:
Pharmacodynamics in terms of platelet reactivity as measured by P2Y12 Reaction Units (PRU) using VerifyNow™ after loading dose of Ticagrelor | Predose, 0h, 2h,6h,12h,24h,36h,48h,60h,72h,84h and 96h
Pharmacodynamics in terms of platelet reactivity as measured by P2Y12 Reaction Units (PRU) using VerifyNow™ after loading dose of Clopidogrel | Predose, 0h, 2h,6h,12h,24h,36h,48h,60h,72h,84h and 96h
Pharmacodynamics in terms of percent of inhibition of adenosine phosphatase (ADP)-induced platelet aggregation assessed by light transmission aggregometry (LTA) after loading dose of Clopidogrel | Predose, 0h, 2h,6h,12h,24h,36h,48h,60h,72h,84h and 96h
Safety profile in terms of adverse events, blood pressure, pulse, temperature, ECG (Electrocardiogram), physical examination, and safety laboratory variables | up to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Carlson, MD, Study Chair — AstraZeneca Wilmington US; Phil Leese, MD, Principal Investigator — Overland Park US, Quintiles, Inc; Judi Hsia, MD, Study Director — Wilmington, US AstraZeneca
Locations (1):
- Research Site, Overland Park, Kansas, United States